CLINICAL TRIAL: NCT02051088
Title: Swedish Drug-elution Trial in Peripheral Arterial Disease - a Multicenter, Prospective Randomized Controlled Clinical Trial Based on the Swedish Vascular Registry (SWEDVASC) Platform
Brief Title: Swedish Drug-elution Trial in Peripheral Arterial Disease
Acronym: SWEDEPAD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: The Swedish Research Council (Other Government); Swedish Heart Lung Foundation (Other); Uppsala University (Other); The Swedish National Registry for Vascular Surgery (Other)
Responsible Party: Principal Investigator, Mårten Falkenberg, MD, PhD, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SWEDEPAD
Record Dates: First submitted 2014-01-27; First posted 2014-01-31 (Estimated); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Peripheral Arterial Disease; Critical Limb Ischemia; Intermittent Claudication
Keywords: Critical limb ischemia; Intermittent claudication; endovascular treatment; drug-elution
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia; Intermittent Claudication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Revascularization with drug eluting technology (Experimental): Revascularization with drug eluting technology
  Interventions: Procedure: Revascularization with drug-eluting technology; Device: drug-coated balloons and/or drug-eluting stents
- Revascularization without drug elution (Active Comparator): Revascularization without drug elution technology
  Interventions: Procedure: Revascularization without drug-eluting technology

INTERVENTIONS:
Procedure: Revascularization with drug-eluting technology — Endovascular intervention with the use of drug-eluting devices (drug-coated balloons and/or drug-eluting stents).
  Arms: Revascularization with drug eluting technology
Procedure: Revascularization without drug-eluting technology — Endovascular intervention without using drug-eluting balloons or stents
  Arms: Revascularization without drug elution
Device: drug-coated balloons and/or drug-eluting stents
  Arms: Revascularization with drug eluting technology

SUMMARY:
Peripheral arterial disease (PAD) causes reduced blood flow to the lower limb(s) due to stenosis or occlusion in the supplying arteries. Symptoms of PAD range from ischemic rest pain and/or ischemic ulcers/gangrene (critical limb ischemia), putting the extremity at risk of amputation, to exercise-induced pain (intermittent claudication), limiting the patients daily activities. Invasive treatments are often indicated to prevent amputations and to alleviate symptoms. More than two thirds of these procedures are presently performed with endovascular techniques (i.e. percutaneous transluminal angioplasty, PTA with or without stent implantation).

In coronary artery disease, stents eluting anti-proliferative drugs (drug eluting stents, DES) reduce restenosis and improve clinical results for the majority of patients. Drug eluting balloons (DEB) are a promising alternative, but there is still little evidence that DES or DEB technology improve clinical outcome in PAD. However, promising results utilizing these new technologies in PAD have been reported in a few studies.

In this trial, we test the hypothesis that drug eluting (DE) technology is superior to conventional endovascular treatment (no-DE) in terms of important clinical outcomes, when applied on infrainguinal (femoropopliteal and/or infrapopliteal) obstructive vascular lesions. The trial consists of 2 separate parallel studies, SWEDEPAD 1 and SWEDEPAD 2, each defined by the severity of peripheral arterial disease. Patients with critical limb ischemia are allocated to SWEDEPAD 1 and patients with intermittent claudication are allocated to SWEDEPAD 2.

ELIGIBILITY:
Inclusion Criteria:

* All adults > 18 years old willing to be randomized
* Symptomatic PAD (critical limb ischemia or intermittent claudication) caused by >50% stenosis or occlusion of infrainguinal arteries and eligible for endovascular treatment according to established indications

Exclusion Criteria:

* Acute thromboembolic disease in the leg
* Infrainguinal aneurysmal disease
* Previous participation in the study or in other randomised interventional study of infrainguinal lesions
* Patients without a Swedish personal identification number

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3556 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Amputation rate (SWEDEPAD 1) | Assessed when all patients have been followed for at least one year
  Primary endpoint for patients with critical limb ischemia (SWEDEPAD 1) is amputation rate during follow-up, analysed when all patients have been followed for at least one year.
Health-related quality of life (SWEDEPAD 2) | Assessed one year after randomization
  Primary endpoint for patients with intermittent claudication (SWEDEPAD 2) is health-related quality of life after one year, assessed with VascuQol-6, a disease-specific health related quality of life instrument in PAD.

SECONDARY OUTCOMES:
Amputation-free survival | Assessed when all participants have been followed for at least one, three and five years.
Survival | Assessed when all participants have been followed for at least one, three and five years.
Target lesion revascularization (TLR) | Assessed one year after the intervention and when all participants have been followed for one, three and five years.
  Need for re-intervention during follow-up
Time to target lesion revascularization | Assessed one year after the intervention and when all participants have been followed for one, three and five years.
Patency | Assessed after 1 month and 1 year
  Patency, defined as freedom from binary restenosis, a reduction in lumen diameter ≥50% in patients assessed with duplex ultrasound after one month and after one year (only certain centres).
Improvement in clinical symptoms, assessed with the Rutherford classification | Assessed after one month and one year
  Particularly changes from Rutherford categories 4, 5 and 6 to lower categories will analysed (SWEDEPAD 1)
  Particularly changes from Rutherford categories 2 and 3 to other categories will analysed (SWEDEPAD 2)
Health-related quality of life (SWEDEPAD 1) | Assessed after one year following randomisation
  Health-related quality of life, assessed with the disease-specific instrument VascuQoL-6
Amputation rate (SWEDEPAD 2) | Assessed one year after the intervention and when all participants have been followed for one, three and five years
Health-economic assessment | Assessed one year after the intervention and when all participants have been followed for one, three and five years
  Assessment of cost-effectiveness and clinical utility (only certain centres).

CONTACTS AND LOCATIONS:
Overall Officials: Mårten Falkenberg, MD, PhD, Principal Investigator — Department of Radiology, Sahlgrenska University Hospital; Joakim Nordanstig, MD, Study Chair — Department of Vascular Surgery, Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Falkenberg M, James S, Andersson M, Andersson M, Delle M, Engstrom J, Fransson T, Gillgren P, Hilbertson A, Horer TM, Jacobsson E, Kragsterman B, Lindback J, Lindgren H, Ludwigs K, Mellander S, Nelzen O, Olin R, Sigvant B, Skoog P, Starck J, Tegler G, Thorbjornsen K, Truedson M, Wahlgren CM, Wallinder J, Ojersjo A, Nordanstig J; SWEDEPAD trial investigators. Paclitaxel-coated versus uncoated devices for infrainguinal endovascular revascularisation in chronic limb-threatening ischaemia (SWEDEPAD 1): a multicentre, participant-masked, registry-based, randomised controlled trial. Lancet. 2025 Sep 13;406(10508):1103-1114. doi: 10.1016/S0140-6736(25)01585-5. Epub 2025 Aug 31. PMID 40902617
- [Derived] Nordanstig J, James S, Andersson M, Andersson M, Delle M, Engstrom J, Fransson T, Gillgren P, Hilbertson A, Horer TM, Jacobsson E, Kragsterman B, Lindback J, Lindgren H, Ludwigs K, Mellander S, Nelzen O, Olin R, Sigvant B, Skoog P, Starck J, Tegler G, Thorbjornsen K, Truedson M, Wahlgren CM, Wallinder J, Ojersjo A, Falkenberg M; SWEDEPAD trial investigators. Paclitaxel-coated versus uncoated devices for infrainguinal endovascular revascularisation in patients with intermittent claudication (SWEDEPAD 2): a multicentre, participant-masked, registry-based, randomised controlled trial. Lancet. 2025 Sep 13;406(10508):1115-1127. doi: 10.1016/S0140-6736(25)01584-3. Epub 2025 Aug 31. PMID 40902614
- [Derived] Nordanstig J, James S, Andersson M, Andersson M, Danielsson P, Gillgren P, Delle M, Engstrom J, Fransson T, Hamoud M, Hilbertson A, Johansson P, Karlsson L, Kragsterman B, Lindgren H, Ludwigs K, Mellander S, Nyman N, Renlund H, Sigvant B, Skoog P, Starck J, Tegler G, Toivola A, Truedson M, Wahlgren CM, Wallinder J, Ojersjo A, Falkenberg M. Mortality with Paclitaxel-Coated Devices in Peripheral Artery Disease. N Engl J Med. 2020 Dec 24;383(26):2538-2546. doi: 10.1056/NEJMoa2005206. Epub 2020 Dec 9. PMID 33296560